CLINICAL TRIAL: NCT05222113
Title: OBSERVATIONAL STUDY OF COMPARISON EFFECTIVITY BETWEEN REMDESIVIR AND FAVIPIRAVIR IN SURABAYA, INDONESIA
Status: Completed | Type: Observational
Sponsor: Bernadette Dian Novita, MD.,PhD (Other)
Responsible Party: Sponsor-Investigator, Bernadette Dian Novita, MD.,PhD, MD.,PhD, Universitas Katolik Widya Mandala Surabaya
Organization: Universitas Katolik Widya Mandala Surabaya (Other)
Other Study IDs: 148/WM12/KEPK/MHSW
Record Dates: First submitted 2022-01-23; First posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Duration of Hospitalization; Clinical Manifestation of COVID-19
MeSH Terms: interventions — remdesivir; favipiravir

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Remdesivir — The patients, based on their clinical condition, got remdesivir OR favipiravir at least five days of treatment. The WHO ordinal scale was used to assess patients' clinical progress in the first and second weeks.
  Other Names: Favipiravir

SUMMARY:
In order to compare the effectiveness between Remdesivir and Favipiravir, an observational analytic study using a retrospective cohort design. Eighty-eight medical records of COVID-19 patients from January to August 2021

DETAILED DESCRIPTION:
Coronavirus Disease 2019 (COVID-19) is an infectious disease caused by Severe Acute Respiratory Syndrome Coronavirus 2 (SARS CoV-2). Antiviral therapies are considered to be one of the COVID-19 treatments. Remdesivir and favipiravir are the antivirals recommended by Indonesia's 3rd COVID-19 Management Guidelines. They have a similar mechanism to inhibit virus replication, specifically by inhibiting RNA-dependent RNA polymerase (RdRp) of the virus. Several studies reported that patients who received these antivirals had a lower duration of hospitalization. However, the effectiveness comparison of remdesivir and favipiravir remains unknown.

An observational analytic study using a retrospective cohort design. Eighty-eight medical records of COVID-19 patients from January to August 2021 are collected by consecutive sampling technique, and this research was carried out at Gotong Royong Hospital Surabaya.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (eighteen years old or above) with moderate to severe COVID-19 (categorized based on KEPUTUSAN MENTERI KESEHATAN REPUBLIK INDONESIA NOMOR HK. 01. 07/MENKES/413/2020);
* Admitted to Gotong Royong Hospital Surabaya from January 2021 to August 2021;
* Received remdesivir OR favipiravir with minimal five days of treatment
* Not in pregnancy and lactating condition

Exclusion Criteria:

* female patient with pregnancy and lactation
* patient whom was passed away or forced home during two-weeks observation period

Ages: 18 Years to 97 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients' medical records from Gotong Royong Surabaya Hospital were obtained from January 2021 to March 2021 and June 2021 to August 2021, since remdesivir was rarely used from April 2021 to May 2021.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-09-25 (Actual); Study Completion 2021-09-25 (Actual)

PRIMARY OUTCOMES:
Clinical manifestation | 2 weeks since drug (remdesivir OR favipiravir) administration
  Oxygen needs, cough, dyspnea

CONTACTS AND LOCATIONS:
Locations (1):
- Gotong Royong Surabaya Hospital, Surabaya, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP